CLINICAL TRIAL: NCT05786742
Title: ULTRA-HYPO Fractionated (UHF) Compared to Moderate-HYPO Fractionated (MHF) Prostate IGRT With HDR Brachytherapy BOOST : A Phase 1-2 Study.
Brief Title: Ultra Hypofractionnated Radiotherapy With HDR Brachytherapy Boost.
Acronym: HYPO-5
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Principal Investigator, André-Guy Martin, Clinical professor, M.D., M.Sc., F.R.C.P.C., CHU de Quebec-Universite Laval
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYPO-5
Record Dates: First submitted 2022-12-23; First posted 2023-03-28 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer; Radiotherapy Side Effect; Hypofractionation; Brachytherapy; Radiotherapy; Localized Prostate Carcinoma
Keywords: hypo fractionation; brachytherapy; Ultra Hypo fractionation
MeSH Terms: conditions — Prostatic Neoplasms; Radiation Injuries

STUDY DESIGN:
Intervention Model Description: Prospective comparative cohort study with non inferiority analysis UH-IMRT combined to 15 Gy HDR Brachytherapy will considerably reduce the treatment fraction delivered while maintaining b-DFS and Side-effects at comparable levels to our actual reported prostate cancer patient population, without lymph nodes involvement (risk being less than 15%). We believe that this therapeutic regime will show to be non-inferior to our actual standard therapeutic regime
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultra hypo fractionation radiation therapy (Experimental): comparative PRO's of 25 Gy in 5 daily fractions (Ultra hypo fractionation) administered to prostate and 1st centimeter of proximal seminal vesicle, starting mid week and ending mid following week.
  Interventions: Radiation: grade and compare reported side effects between groups
- moderate hypo fractionation radiation therapy (Active Comparator): PRO's of moderate hypo fractionation, 37,5 Gy in 15 or 36 Gy in 12 daily fractions administered 5 days per week.
  Interventions: Radiation: grade and compare reported side effects between groups

INTERVENTIONS:
Radiation: grade and compare reported side effects between groups — Compare experimental ultra hypo fractionation (25 Gy in 5 daily fractions administered starting mid week and ending mid following week) to our standard fractionation (either 37,5 Gy given in 15 daily fractions, or 36 Gy in 12 daily fractions).
  * Toxicity analysis will be quantitatively evaluated using CTCAE (v5) at 1, 2 and 5 years post-therapy, and has needed at FU visits. Kaplan-Meier statistical analysis will be used to report toxicity evolution through time.
  * median IPSS scores will be reported at 3, 6, 12 months and yearly (1, 2, 3, 4 et 5) post-therapy. IPSS median time to baseline return will be calculated.
  * IPSS urinary scores, sexual function (SHIM) and GI toxicity (CTCAE-v5) and quality of life questionnaires ( EPIC-26) will be given at 3, 6 months and yearly thereafter (1, 2, 3, 4 et 5) post-treatment.
  Other Names: report and compare IPSS scores; report and compare EPIC26 scores; report and compare SHIM scores; report and compare CTCAE scores; report and compare clinical outcomes

SUMMARY:
Phase 1-2 study, comparing ultra-hypofractionnated (UH) to a moderately hypofractionnated (MH) radiation therapy, with image guided HDR prostate brachytherapy. Using iso-equivalent doses, a non-inferiority analysis will be done in order to prove UH non-inferior to MH, toxicity wise. Acceptability, tolerability, acute and late toxicity will be reported. MRI visible dominant intra-prostatic lesion will be outlines and variability between radiation oncologists and radiologists will be reported. As secondary objective, biochemical and clinical failure free survival will be reported at 5 & 10 years.

DETAILED DESCRIPTION:
Phase 1 : consists in a feasibility study (First 28 patients).

Phase 2 : monocentric prospective comparative cohort study.

Recruitment :

* "Centre intégré de cancérologie du CHU de Québec-Université Laval."
* Recruitment period: December 2015 to June 2023

Brachytherapy :

* Implantation under general or spinal anesthesia
* Foley catheter insertion in bladder.
* TRUS prostate localisation.
* Prostate volume measurement.
* Gold fiducial markers (3) insertion.
* Prostate brachytherapy catheters (14 à 21) insertion.
* Cystoscopy for bladder and urethra integrity control.
* Re-insertion of foley catheter after cystoscopy.

Planning imaging: TRUS or CT scan (has needed).

Structures delineation by radiation oncologist (brachytherapist).

* Prostate
* Seminale vesicles
* Rectum
* Colon sigmoïde
* Bladder
* Urethra
* Penile bulb

Dosimetric optimisation

* Oncentra Prostate v. 4.2.2 d'Elekta brachytherapy (Veenendaal, The Netherlands)
* Oncentra Brachy version 4.6 (if under CT scan).

Treatment (brachytherapy dose delivery).

* 15 Gy in one fraction
* Direct interstitial dose monitoring (20 patients or more). Fiber-optic dosimeter inserted in prostate brachytherpy catheter for live dose delivery mesurements.

Foley ablation under full bladder, same day or day after therapy.

Radiotherapy:

* Via IMRT, VMAT or SBRT technics.
* Dose : 25 Gy in 5 fractions administered over a 7 days period. 2 to 3 fractions separated by 2 days, weekend break.
* PTV includes prostate and the first centimeter of seminal vesicle.

Simulation

* one week post brachytherapy
* standard has described in the department procedure manual.
* maximal CT scan slice thickness : 2-3mm.
* uretro-graphy done to identify urogenital sphincter.

Multiparametric MRI

* If no counter-indication and available,
* a T2 tridimensional sequence for prostate delineation
* slice thickness : 1 mm.
* a diffusion weighted sequence will be done.
* a DTI with tractography can be done optionally.
* contrast media (gadolinium) is optional.

Physique

* Linac energy (between 6 MV to 18 MV).
* ARC therapy technique will be used
* planification softwares: Éclipse, Pinnacle or Raystation.
* Portal (kV-kV) imagery will be used for marker match.
* CBCT will be done at each fraction delivered.

Clinical and dosimetric data will be collected prior treatment.

Primary objectives :

* Toxicity analysis will be quantitatively evaluated using CTCAE (v5) at 1, 2 and 5 years post-therapy, and has needed at FU visits. Kaplan-Meier statistical analysis will be used to report toxicity evolution through time.
* median IPSS scores will be reported at 3, 6, 12 months and yearly (1, 2, 3, 4 et 5) post-therapy. IPSS median time to baseline return will be calculated.
* IPSS urinary scores, sexual function (SHIM) and GI toxicity (CTCAE-v5) and quality of life questionnaires ( EPIC-26) will be given at 3, 6 months and yearly thereafter (1, 2, 3, 4 et 5) post-treatment.

Secondary objectives : Biochemical disease-free survival has per Phoenix definition (by American Society of Radiation Oncology - ASTRO) recommendation will be reported using Kaplan-Meier analysis.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven Prostate adenocarcinoma
* Stage T1c, T2 (Annex 2)
* Stage Nx or N0
* Stage Mx or M0
* PSA < 20ng/ml
* Gleason Score 6 or 7
* Having the ability to sing a written consent

Exclusion Criteria:

* Age < 18ans
* Clinical Stage T3 or T4
* Stage N1
* Stage M1
* PSA > 20
* Gleason Score 8 to 10
* IPSS Score > 20 alpha-blocking medication.
* Prior pelvic radiotherapy.
* History of active collagenosis (Lupus, Sclerodermia, Dermatomyosis)
* Past history of Inflammatory Bowell Disease
* Bilateral hip prosthesis

Ages: 18 Years to 95 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — men
Enrollment: 205 (Estimated)
Dates: Start 2014-04 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
GU toxicity analysis (CTCAE) | at baseline, prior treatment
  quantitatively evaluated using CTCAE (v5) and compare between arms
GU toxicity analysis (CTCAE) | at 3 months post-therapy
  quantitatively evaluated using CTCAE (v5) and compare between arms
GU toxicity analysis (CTCAE) | at 6 months post-therapy
  quantitatively evaluated using CTCAE (v5) and compare between arms
GU toxicity analysis (CTCAE) | at 1 year post-therapy
  quantitatively evaluated using CTCAE (v5) and compare between arms
GU toxicity analysis (CTCAE) | at 2 years post-therapy
  quantitatively evaluated using CTCAE (v5) and compare between arms
GU toxicity analysis (CTCAE) | at 3 years post-therapy
  quantitatively evaluated using CTCAE (v5) and compare between arms
GU toxicity analysis (CTCAE) | at 4 years post-therapy
  quantitatively evaluated using CTCAE (v5) and compare between arms
GU toxicity analysis (CTCAE) | at 5 years post-therapy
  quantitatively evaluated using CTCAE (v5) and compare between arms
GI toxicity analysis (CTCAE) | at baseline, prior treatment
  quantitatively evaluated using CTCAE (v5) and compare between arms
GI toxicity analysis (CTCAE) | at 3 months post-therapy
  quantitatively evaluated using CTCAE (v5) and compare between arms
GI toxicity analysis (CTCAE) | at 6 months post-therapy
  quantitatively evaluated using CTCAE (v5) and compare between arms
GI toxicity analysis (CTCAE) | at 1 year post-therapy
  quantitatively evaluated using CTCAE (v5) and compare between arms
GI toxicity analysis (CTCAE) | at 2 years post-therapy
  quantitatively evaluated using CTCAE (v5) and compare between arms
GI toxicity analysis (CTCAE) | at 3 years post-therapy
  quantitatively evaluated using CTCAE (v5) and compare between arms
GI toxicity analysis (CTCAE) | at 4 years post-therapy
  quantitatively evaluated using CTCAE (v5) and compare between arms
GI toxicity analysis (CTCAE) | at 5 years post-therapy
  quantitatively evaluated using CTCAE (v5) and compare between arms
urinary toxicity analysis (IPSS) | at baseline, prior treatment
  median IPSS scores will be reported post-therapy and compare between arms at baseline, prior treatment
urinary toxicity analysis (IPSS) | at 3 months
  median IPSS scores will be reported post-therapy and compare between arms at 3 months post-therapy
urinary toxicity analysis (IPSS) | at 6 months
  median IPSS scores will be reported post-therapy and compare between arms at 6 months post-therapy
urinary toxicity analysis (IPSS) | at 1 year
  median IPSS scores will be reported post-therapy and compare between arms at 1 year post-therapy
urinary toxicity analysis (IPSS) | at 2 years
  median IPSS scores will be reported post-therapy and compare between arms at 2 years post-therapy
urinary toxicity analysis (IPSS) | at 3 years
  median IPSS scores will be reported post-therapy and compare between arms at 3 years post-therapy
urinary toxicity analysis (IPSS) | at 4 years
  median IPSS scores will be reported post-therapy and compare between arms at 4 years post-therapy
urinary toxicity analysis (IPSS) | at 5 years
  median IPSS scores will be reported post-therapy and compare between arms at 5 years post-therapy
quality of life questionnaires analysis (EPIC26) | baseline, prior treatment
  median EPIC26 scores will be reported post-therapy and compare between arms at baseline, prior treatment
quality of life questionnaires analysis (EPIC26) | at 3 months
  median EPIC26 scores will be reported post-therapy and compare between arms at 3 months post-treatment
quality of life questionnaires analysis (EPIC26) | at 6 months
  median EPIC26 scores will be reported post-therapy and compare between arms at 6 months post-treatment
quality of life questionnaires analysis (EPIC26) | at 1 year
  median EPIC26 scores will be reported post-therapy and compare between arms at 1 year post-treatment
quality of life questionnaires analysis (EPIC26) | at 2 years
  median EPIC26 scores will be reported post-therapy and compare between arms at 2 years post-treatment
quality of life questionnaires analysis (EPIC26) | at 3 years
  median EPIC26 scores will be reported post-therapy and compare between arms at 3 years post-treatment
quality of life questionnaires analysis (EPIC26) | at 4 years
  median EPIC26 scores will be reported post-therapy and compare between arms at 4 years post-treatment
quality of life questionnaires analysis (EPIC26) | at 5 years
  median EPIC26 scores will be reported post-therapy and compare between arms at 5 years post-treatment
sexual function analysis (SHIM) | baseline, prior treatment
  median SHIM scores will be reported at baseline prior treatment
sexual function analysis (SHIM) | at 3 months
  median SHIM scores will be reported post-therapy and compare between arms at 3 months post-treatment
sexual function analysis (SHIM) | at 6 months
  median SHIM scores will be reported post-therapy and compare between arms at 6 months post-treatment
sexual function analysis (SHIM) | at 1 year
  median SHIM scores will be reported post-therapy and compare between arms at 1 year post-treatment
sexual function analysis (SHIM) | at 2 years
  median SHIM scores will be reported post-therapy and compare between arms at 2 years post-treatment
sexual function analysis (SHIM) | at 3 years
  median SHIM scores will be reported post-therapy and compare between arms at 3 years post-treatment
sexual function analysis (SHIM) | at 4 years
  median SHIM scores will be reported post-therapy and compare between arms at 4 years post-treatment
sexual function analysis (SHIM) | at 5 years
  median SHIM scores will be reported post-therapy and compare between arms at 5 years post-treatment

SECONDARY OUTCOMES:
Clinical outcomes | at 5 years
  Biochemical disease-free survival has per Phoenix definition (by American Society of Radiation Oncology - ASTRO) will be reported using Kaplan-Meier analysis, as well for disease free survival, metastasis free survival and overall survival.
Clinical outcomes | at 10 years
  Biochemical disease-free survival has per Phoenix definition (by American Society of Radiation Oncology - ASTRO) will be reported using Kaplan-Meier analysis, as well for disease free survival, metastasis free survival and overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Andre-Guy Martin, Study Chair — CHU de Québec
Locations (1):
- CHUdeQuebec, Québec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Crook JM, Gomez-Iturriaga A, Wallace K, Ma C, Fung S, Alibhai S, Jewett M, Fleshner N. Comparison of health-related quality of life 5 years after SPIRIT: Surgical Prostatectomy Versus Interstitial Radiation Intervention Trial. J Clin Oncol. 2011 Feb 1;29(4):362-8. doi: 10.1200/JCO.2010.31.7305. Epub 2010 Dec 13. PMID 21149658
- [Result] Bachand F, Martin AG, Beaulieu L, Harel F, Vigneault E. An eight-year experience of HDR brachytherapy boost for localized prostate cancer: biopsy and PSA outcome. Int J Radiat Oncol Biol Phys. 2009 Mar 1;73(3):679-84. doi: 10.1016/j.ijrobp.2008.05.003. Epub 2008 Oct 27. PMID 18963537
- [Result] Grimm P, Billiet I, Bostwick D, Dicker AP, Frank S, Immerzeel J, Keyes M, Kupelian P, Lee WR, Machtens S, Mayadev J, Moran BJ, Merrick G, Millar J, Roach M, Stock R, Shinohara K, Scholz M, Weber E, Zietman A, Zelefsky M, Wong J, Wentworth S, Vera R, Langley S. Comparative analysis of prostate-specific antigen free survival outcomes for patients with low, intermediate and high risk prostate cancer treatment by radical therapy. Results from the Prostate Cancer Results Study Group. BJU Int. 2012 Feb;109 Suppl 1:22-9. doi: 10.1111/j.1464-410X.2011.10827.x. PMID 22239226
- [Result] Morris WJ, Keyes M, Palma D, Spadinger I, McKenzie MR, Agranovich A, Pickles T, Liu M, Kwan W, Wu J, Berthelet E, Pai H. Population-based study of biochemical and survival outcomes after permanent 125I brachytherapy for low- and intermediate-risk prostate cancer. Urology. 2009 Apr;73(4):860-5; discussion 865-7. doi: 10.1016/j.urology.2008.07.064. Epub 2009 Jan 24. PMID 19168203
- [Result] Morris WJ, Keyes M, Spadinger I, Kwan W, Liu M, McKenzie M, Pai H, Pickles T, Tyldesley S. Population-based 10-year oncologic outcomes after low-dose-rate brachytherapy for low-risk and intermediate-risk prostate cancer. Cancer. 2013 Apr 15;119(8):1537-46. doi: 10.1002/cncr.27911. Epub 2012 Dec 26. PMID 23280183
- [Result] Morton G, Loblaw A, Cheung P, Szumacher E, Chahal M, Danjoux C, Chung HT, Deabreu A, Mamedov A, Zhang L, Sankreacha R, Vigneault E, Springer C. Is single fraction 15 Gy the preferred high dose-rate brachytherapy boost dose for prostate cancer? Radiother Oncol. 2011 Sep;100(3):463-7. doi: 10.1016/j.radonc.2011.08.022. Epub 2011 Sep 14. PMID 21924511
- [Result] Wright JL, Izard JP, Lin DW. Surgical management of prostate cancer. Hematol Oncol Clin North Am. 2013 Dec;27(6):1111-35, vii. doi: 10.1016/j.hoc.2013.08.010. PMID 24188255
- [Result] Stone NN, Stock RG, Cesaretti JA, Unger P. Local control following permanent prostate brachytherapy: effect of high biologically effective dose on biopsy results and oncologic outcomes. Int J Radiat Oncol Biol Phys. 2010 Feb 1;76(2):355-60. doi: 10.1016/j.ijrobp.2009.01.078. Epub 2009 Jul 23. PMID 19632069
- [Result] Viani GA, Stefano EJ, Afonso SL. Higher-than-conventional radiation doses in localized prostate cancer treatment: a meta-analysis of randomized, controlled trials. Int J Radiat Oncol Biol Phys. 2009 Aug 1;74(5):1405-18. doi: 10.1016/j.ijrobp.2008.10.091. PMID 19616743
- [Result] Holm HH, Gammelgaard J. Ultrasonically guided precise needle placement in the prostate and the seminal vesicles. J Urol. 1981 Mar;125(3):385-7. doi: 10.1016/s0022-5347(17)55044-2. No abstract available. PMID 7206090
- [Result] Hill RP, Rodemann HP, Hendry JH, Roberts SA, Anscher MS. Normal tissue radiobiology: from the laboratory to the clinic. Int J Radiat Oncol Biol Phys. 2001 Feb 1;49(2):353-65. doi: 10.1016/s0360-3016(00)01484-x. PMID 11173128
- [Result] Williams MV, Denekamp J, Fowler JF. A review of alpha/beta ratios for experimental tumors: implications for clinical studies of altered fractionation. Int J Radiat Oncol Biol Phys. 1985 Jan;11(1):87-96. doi: 10.1016/0360-3016(85)90366-9. PMID 3881377
- [Result] McCammon R, Rusthoven KE, Kavanagh B, Newell S, Newman F, Raben D. Toxicity assessment of pelvic intensity-modulated radiotherapy with hypofractionated simultaneous integrated boost to prostate for intermediate- and high-risk prostate cancer. Int J Radiat Oncol Biol Phys. 2009 Oct 1;75(2):413-20. doi: 10.1016/j.ijrobp.2008.10.050. Epub 2009 Apr 11. PMID 19362783
- [Result] Schmidt MA, Payne GS. Radiotherapy planning using MRI. Phys Med Biol. 2015 Nov 21;60(22):R323-61. doi: 10.1088/0031-9155/60/22/R323. Epub 2015 Oct 28. PMID 26509844
- [Result] Arcangeli G, Saracino B, Gomellini S, Petrongari MG, Arcangeli S, Sentinelli S, Marzi S, Landoni V, Fowler J, Strigari L. A prospective phase III randomized trial of hypofractionation versus conventional fractionation in patients with high-risk prostate cancer. Int J Radiat Oncol Biol Phys. 2010 Sep 1;78(1):11-8. doi: 10.1016/j.ijrobp.2009.07.1691. Epub 2010 Jan 4. PMID 20047800
- [Result] D'Amico AV, Chen MH, Renshaw AA, Loffredo M, Kantoff PW. Androgen suppression and radiation vs radiation alone for prostate cancer: a randomized trial. JAMA. 2008 Jan 23;299(3):289-95. doi: 10.1001/jama.299.3.289. PMID 18212313
- [Result] Jones CU, Hunt D, McGowan DG, Amin MB, Chetner MP, Bruner DW, Leibenhaut MH, Husain SM, Rotman M, Souhami L, Sandler HM, Shipley WU. Radiotherapy and short-term androgen deprivation for localized prostate cancer. N Engl J Med. 2011 Jul 14;365(2):107-18. doi: 10.1056/NEJMoa1012348. PMID 21751904
- [Result] Partin AW, Mangold LA, Lamm DM, Walsh PC, Epstein JI, Pearson JD. Contemporary update of prostate cancer staging nomograms (Partin Tables) for the new millennium. Urology. 2001 Dec;58(6):843-8. doi: 10.1016/s0090-4295(01)01441-8. PMID 11744442
- [Result] Gregoire JP, Moisan J, Labrecque M, Cusan L, Diamond P. [Validation of a French adaptation of the international prostatic symptom score]. Prog Urol. 1996 Apr;6(2):240-9. French. PMID 8777417